CLINICAL TRIAL: NCT04280887
Title: MyPad - Intelligent Bladder Pre-void Alerting System
Acronym: MyPad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Central Lancashire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: My Pad Protocol version 1
Record Dates: First submitted 2020-02-05; First posted 2020-02-21 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Enuresis, Nocturnal; Enuresis
MeSH Terms: conditions — Nocturnal Enuresis; Enuresis

STUDY DESIGN:
Intervention Model Description: Cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will wear the device for the specified test period (3 months)
  Interventions: Device: MyPad

INTERVENTIONS:
Device: MyPad — Ultrasound bed wetting alarm

SUMMARY:
Development a 'dry alarm' that can help children and adolescents become dry at night.

DETAILED DESCRIPTION:
Enuresis / Bedwetting is a common problem causing much emotional distress. Most children are dry by the age of 5 years, but a significant number of older children still wet their bed. This can be very distressing for child and family. There is also an associated cost due to extra laundry and impact of lost sleep.

Programmes to help children become dry at night often include the use of a moisture alarm. The alarms sound when the child begins to wet the bed, waking them up to go to the toilet instead. Most alarms work by detecting wetness, sounding the alarm when the child starts to pass urine. As such, they still need to change pyjamas and bed sheets.

The investigators aim to develop a 'dry alarm' that can help children and adolescents become dry at night. The alarm will sound when the bladder is full, before the child passes urine. This would avoid wet beds. The investigators have engineered parts for this alarm, but need to work on making it ready for use. This device will enable children to have dry nights whilst learning bladder control.

This study has several phases. The alarm will consist of a small box worn over the abdomen. The aim is to test this overnight, and adjust it for comfort and ease. The device uses a mini ultrasound machine, which measures how much urine is in the bladder. There will be a series of tests to calibrate the device compared to a clinical ultrasound device. Then children with enuresis/ bed wetting will wear it overnight. It will be linked to an alarm which will sound once the bladder is full.

This particular study will determine the feasibility of the product, to confirm the design and specifications, including a comfort trial, calibration and comparison with clinical scans, and operating process prior to a future clinical trial.

The total number of participants is 25 - however this will be split over the different phases of the trial.

Comfort Trial - 5 Calibration trial 3 month testing phase - 10

ELIGIBILITY:
Inclusion Criteria:

* Age 7 years to 12 years
* Bedwetting twice a week or more
* Good understanding of English language
* For the initial comfort trials and the calibration trial healthy volunteers may be invited to take part.

Exclusion Criteria:

* there is a medical cause for bedwetting
* they have significant learning difficulties
* they are obese (above 98th centile for Body Mass Index)
* they have severe hearing impairment

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Bladder expansion | 3 months
  Bladder size measurements, device is able to provide consistent readings
Reduction in adverse events | 3 months
  Number of adverse events measured over the three months - reduction over time

SECONDARY OUTCOMES:
Comfort | 3 months
  Comfort, design and tolerability of device using validated comfort tool

CONTACTS AND LOCATIONS:
Locations (1):
- Lancashire Teaching Hospitals NHS Foundation Trust, Preston, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT04280887/Prot_000.pdf